CLINICAL TRIAL: NCT01827566
Title: Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial With a Cross-over Design to Assess the Prevalence of Non Celiac Gluten Sensitivity Among Patients Spontaneously Adherent to Gluten Free Diet
Brief Title: Prevalence of Non Celiac Gluten Sensitivity Among Patients Spontaneously Adherent to Gluten Free Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Alberto Lanzini, MD PhD, Associate Professor of Gastroenterology, Università degli Studi di Brescia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE-2012-GS
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Non Celiac Gluten Sensitivity
Keywords: Celiac Disease; Gluten Sensitivity; Gluten; Double-blind challenge, placebo-controlled challenge; Gluten free flour
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- gluten (Active Comparator): 10 grams of gluten in each sachet to be dispersed daily on food for ten days, while maintaining a gluten free diet
  Interventions: Other: gluten
- gluten free flour (Placebo Comparator): 10 grams of gluten free flour in each sachet to be dispersed daily on food for ten days, while maintaining a gluten free diet
  Interventions: Other: gluten free flour

INTERVENTIONS:
Other: gluten
  Arms: gluten
Other: gluten free flour
  Arms: gluten free flour

SUMMARY:
The purpose of this study is to assess the prevalence of Gluten Sensitivity, by a double-blind placebo-controlled challenge with gluten, followed by two months period of Low-FODMAPs (Fermentable Oligosaccharides Disaccharides Monosaccharides And Polyols) diet, in patients spontaneously adherent to gluten free diet because of symptoms upon gluten exposure and in whom diagnosis of Celiac Disease and Wheat Allergy has been ruled out.

ELIGIBILITY:
Inclusion Criteria:

* Adherence to gluten free diet without medical need
* Negative Celiac Disease related serology (while on gluten containing diet)
* Normal villous structure at duodenal biopsy (while on gluten containing diet)

Exclusion Criteria:

* Diagnosis of Celiac Disease
* Diagnosis of Wheat Allergy
* Diagnosis of organic gastrointestinal disease
* Severe concomitant disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Patient's ability to correctly identify the phase with gluten | Time (days) 35
  * time 0: start of first challenge (phase A, either with gluten or gluten free flour)
  * time 10: end of phase A and start of wash-out period
  * time 25: end of wash-out period and start of second challenge (phase B, either with gluten or gluten free flour)
  * time 35: end of phase B

SECONDARY OUTCOMES:
Changes in serum level of anti-tissue transglutaminases immunoglobulin A (IgA)/immunoglobulin G (IgG) and of anti-gliadin IgA/IgG | Time (days) 0, 10, 25, 35
  * time 0: start of first challenge (phase A, either with gluten or gluten free flour)
  * time 10: end of phase A and start of wash-out period
  * time 25: end of wash-out period and start of second challenge (phase B, either with gluten or gluten free flour)
  * time 35: end of phase B
Change in Fatigue Visual Scale | Time (days) 0, 10, 25, 35
  * time 0: start of first challenge (phase A, either with gluten or gluten free flour)
  * time 10: end of phase A and start of wash-out period
  * time 25: end of wash-out period and start of second challenge (phase B, either with gluten or gluten free flour)
  * time 35: end of phase B
Change in Gastrointestinal Rating Score (GSRS) during Challenge with and without gluten | Time (days) 0,10, 25, 35
  * Time 0: Start of first challenge (phase A, either with gluten or gluten free flour)
  * Time 10: end of phase A and start of wash-out period
  * Time 25: end of wash-out period and start of second challenge (phase B, either with gluten or gluten free flour)
  * Time 35: end of phase B
  * At the beginning of Low-FODMAPs diet
  * After two months of Low-FODMAPs diet
Change in symptoms' score (1 to 7 Likert scale) as recorded on a daily diary | From Time 0 (days) to 10 and from 25 to 35
  * time 0: start of first challenge (phase A, either with gluten or gluten free flour)
  * time 10: end of phase A and start of wash-out period
  * time 25: end of wash-out period and start of second challenge (phase B, either with gluten or gluten free flour)
  * time 35: end of phase B

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Lanzini, MD, PhD, Study Chair — University of Brescia, Unit of Gastroenterology; Barbara Zanini, MD, PhD, Principal Investigator — University of Brescia, Unit of Gastroenterology; Chiara Ricci, MD, PhD, Principal Investigator — University of Brescia, Unit of Gastroenterology
Locations (1):
- University and Spedali Civili of Brescia, Unit of Gastroenterology, Brescia, Italy